## The Safety and Efficacy of the Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) for Short Laryngologic Surgical Procedures

Statistical Analysis Plan
NCT03091179
June 20, 2019

Means and standard deviations were calculated for each of the patient characteristics. The statistical significance of differences between THRIVE and non-THRIVE patients was assessed using a *t*-test for all patient characteristics except gender, where a chi-square text was used. No adjustments were made to the statistical significance threshold for multiple comparisons, and our results should be viewed as exploratory.